CLINICAL TRIAL: NCT02329613
Title: Impact of the Introduction of a New Qualitative Composition of the Evening Meal on the Feeding Behavior of Institutionalized Residents of a Long-term Care Unit: a Randomized, Single Center Study
Brief Title: Introduction of an Enriched Evening Meal on the Feeding Behavior of Institutionalized Residents
Acronym: IRCAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: LOCAL/2014/BH-01; 2014-A00509-38 (Other: RCB number)
Record Dates: First submitted 2014-12-29; First posted 2014-12-31 (Estimated); Last update posted 2016-05-24 (Estimated); Status verified 2016-04

CONDITIONS: Institutionalization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard evening meal (Active Comparator): Patients randomized to this arm will receive standard evening meals.
  Intervention: Standard evening meals.
  Interventions: Other: Standard evening meals.
- Improved evening meal (Experimental): Patients randomized to this arm will receive improved evening meals. Improved meals will include enriched soup (with starches, butter, cheese or sour cream), a semi-liquid dairy dessert, fruit or a fruit dessert.
  Intervention: Improved evening meal
  Interventions: Other: Improved evening meal

INTERVENTIONS:
Other: Standard evening meals. — Patients will receive usual evening meals.
  Arms: Standard evening meal
Other: Improved evening meal — Patients will receive improved evening meals. Improved meals will include enriched soup (with starches, butter, cheese or sour cream), a semi-liquid dairy dessert, fruit or a fruit dessert.
  Arms: Improved evening meal

SUMMARY:
The main objective of this study was to evaluate and compare 6-month calorie intakes between a group of patients receiving a standard dinner and a group of patients whose evening meal is "improved"; compliance will be assessed on a food card with 5 levels of consumption: no (0%), 25%, 50%, 75%, all (100%). This per patient per meal food card will be prepared 3 days per month for 6 months and will, from the total calorie intake of each dish, estimate calorie intake ingested per day on all meals of the day.

DETAILED DESCRIPTION:
The secondary objectives of this study are to evaluate the two groups for the following:

A. The difference between 0 and 6 months in: the patient's weight, calorie intake, serum prealbumin, albumin and CRP, blood sugar for diabetic patients.

B. Monthly evolution over 6 months: calorie intake, the patient's weight. C. The quarterly trend over 6 months: serum prealbumin, albumin and CRP, blood sugar for diabetic patients.

D. Comorbidities and mortality. E. the risk of morning hypoglycaemia for diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* The subject or his/her representative must be given free and informed consent and must have signed the consent
* The subject must be affiliated with or beneficiary of a health insurance plan
* The subject has lived for at least 3 months in the institution
* The subject is fed by mouth only

Exclusion Criteria:

* The subject is participating in another study
* The subject is in an exclusion period determined by a previous study
* The subject or his/her legal representative refuses to sign the consent
* It is not possible to correctly inform the subject or his/her representative

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 48 (Actual)
Dates: Start 2015-04; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Total caloric ration for each dish | 6 months
Meal compliance for 3 days | 6 months
Ingested caloric intake | 6 months

SECONDARY OUTCOMES:
Total caloric ration for each dish | Baseline (days -7 to 0)
Total caloric ration for each dish | Month 1
Total caloric ration for each dish | Month 2
Total caloric ration for each dish | Month 3
Total caloric ration for each dish | Month 4
Total caloric ration for each dish | Month 5
Meal compliance for 3 days | Baseline (days -7 to 0)
Meal compliance for 3 days | Month 1
Meal compliance for 3 days | Month 2
Meal compliance for 3 days | Month 3
Meal compliance for 3 days | Month 4
Meal compliance for 3 days | Month 5
Ingested caloric intake | Baseline (days -7 to 0)
Ingested caloric intake | Month 1
Ingested caloric intake | Month 2
Ingested caloric intake | Month 3
Ingested caloric intake | Month 4
Ingested caloric intake | Month 5
Weight (kg) | Baseline (days -7 to 0)
Weight (kg) | Month 1
Weight (kg) | Month 2
Weight (kg) | Month 3
Weight (kg) | Month 4
Weight (kg) | Month 5
Weight (kg) | Month 6
Serum prealbumin | Baseline (days -7 to 0)
Serum prealbumin | Month 3
Serum prealbumin | Month 6
Serum albumin | Baseline (days -7 to 0)
Serum albumin | Month 3
Serum albumin | Month 6
Serum C reactive protein | Baseline (days -7 to 0)
Serum C reactive protein | Month 3
Serum C reactive protein | Month 6
Glycated hemoglobin (HbA1C) for diabetic patients | Baseline (days -7 to 0)
Glycated hemoglobin (HbA1C) for diabetic patients | Month 3
Glycated hemoglobin (HbA1C) for diabetic patients | Month 6
Presence/absence of comorbidities | Month 6
Mortality | Month 6
Capillary fasting blood glucose for diabetic patients | Month 1
Capillary fasting blood glucose for diabetic patients | Month 2
Capillary fasting blood glucose for diabetic patients | Month 3
Capillary fasting blood glucose for diabetic patients | Month 4
Capillary fasting blood glucose for diabetic patients | Month 5
Capillary fasting blood glucose for diabetic patients | Month 6

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Rouvière, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes; Béatrice Hébert, Nurse, Study Director — Centre Hospitalier Universitaire de Nîmes
Locations (1):
- CHRU de Nîmes - Centre de Gérontologie de Serre Cavalier, Nîmes, France